CLINICAL TRIAL: NCT03261284
Title: D-dimer to Improve Anticoagulation Management in Adult Patients Supported With Extracorporeal Membrane Oxygenation: a Prospective Cohort Study
Brief Title: D-dimer to Improve Anticoagulation Outcome During ECMO loNg-term supporteD
Acronym: DIAMOND
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Wuhan Asia Heart Hospital (Other)
Responsible Party: Principal Investigator, Litao Zhang, Director of Thrombosis centre, Wuhan Asia Heart Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2017-P-032
Record Dates: First submitted 2017-08-22; First posted 2017-08-24 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Extracorporeal Membrane Oxygenation Complication; Thrombosis; Hemorrhage; Heparin Overdose
Keywords: D-dimer; Extracorporeal Membrane Oxygenation; heparin; anticoagulant
MeSH Terms: conditions — Thrombosis; Hemorrhage

STUDY DESIGN:
Intervention Model Description: D-dimer is mornitored. If D-dimer levels continue to rise (>1.5 times previous result ), increase the dose of heparin to reach the upper limit of the treatment target; If the D-dimer levels is stable (<1.5 times previous result ) or is decreasing, the anticoagulation dose is maintained at current level (no active bleeding) or decreased (active bleeding).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DIAMOND group (Experimental): D-dimer and anti-Xa are mornitored. If D-dimer levels continue to rise (>1.5 times previous result ), increase the dose of heparin to reach the upper limit of the treatment target; If the D-dimer levels is stable (<1.5 times previous result ) or is decreasing, the anticoagulation dose is maintained at current level (no active bleeding) or decreased (active bleeding).
  Interventions: Diagnostic Test: D-dimer-guided adjustment stratege
- Control group (Active Comparator): Heparin dose adjusted according to anti-Xa activity or activated partial thromboplastin time (aPTT). The target range is aPTT 1.5 to 2.5 times the upper limit of normal or therapeutic anti-Xa levels (0.3 U/ml to 0.7 U/ml) for unfractionated heparin.
  Interventions: Diagnostic Test: Thepeautic-heparin therapy

INTERVENTIONS:
Diagnostic Test: D-dimer-guided adjustment stratege — D-dimer-guided adjustment stratege
  Other Names: Heparin
  Arms: DIAMOND group
Diagnostic Test: Thepeautic-heparin therapy — 0.3-0.7U/ml of anti-Xa activity or APTT 1.5-2.5 times of control
  Arms: Control group

SUMMARY:
This was a prospective, cohort study.

DETAILED DESCRIPTION:
Adult Patients receiving ECMO surpport in Wuhan Asia Heart Hospital were enrolled by cohort. Unfractionated heparin was used for Anticoagulation therapy, APTT or Anti-Xa activity is monitored for dose adjustment. Meanwhile, D-dimer is mornitored. If D-dimer levels continue to rise (>1.5 times previous result ), increase the dose of heparin to reach the upper limit of the treatment target; If the D-dimer levels is stable (<1.5 times previous result ) or is decreasing, the anticoagulation dose is maintained at current level (no active bleeding) or decreased (active bleeding). All patients were followed up The occurrence of endpoints during in-hospital and 30 days after discharge, including bleeding events, thrombotic events and all-cause deaths were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Adult Patients
* Receiving ECMO surpport for any reason

Exclusion Criteria:

* The duration of ECMO surpport was less than 24 hours .
* Those who had difficulty in compliance or were unavailable for follow-up.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Thrombotic events | 24 months
  Stroke, DVT, PE, Peripheral arterial embolism, ACS etc.
hemorrhagic events | 24 months
  cerebral hemorrhage,Gastrointestinal bleeding etc.

SECONDARY OUTCOMES:
all-cause deaths | 24 months
  all-cause deaths

CONTACTS AND LOCATIONS:
Overall Officials: Zhenlu ZHANG, MD,PhD, Study Director — Wuhan Asia Heart Hospital
Locations (1):
- Zhang litao, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No